CLINICAL TRIAL: NCT04937738
Title: Treatment Discontinuation Associated With Perioperative Toxicity of FLOT Versus XELOX Chemotherapy in Patient With Resectable Gastric Cancer; Phase 2
Brief Title: Perioperative Chemotherapy in Gastric Cancer
Acronym: PECORINO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: High rate of disease progression in XELOX arm
Sponsor: Ukrainian Society of Clinical Oncology (Other)
Responsible Party: Principal Investigator, Oleksii Dobrzhanskiy, Principal investigator, National Cancer Institute (NCI)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 275
Record Dates: First submitted 2021-06-04; First posted 2021-06-24 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Gastric Cancer
Keywords: perioperative chemotherapy; pathological responce rate; gastrectomy; gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; Oxaliplatin; Leucovorin; Fluorouracil; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Perioperative XELOX chemotherapy (Active Comparator): Oxaliplatin 130 mg/m2, d1 Capecitabine 1000 mg/m² two times per day (BID), d1-14, every 3 weeks (q3w) 4 cycles (12 weeks) pre-OP and 3 cycles (12 weeks) post-OP
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin
- Perioperative FLOT chemotherapy (Experimental): Docetaxel 50mg/m2, d1 5-FU 2600 mg/m², d1 Leucovorin 200 mg/m², d1 Oxaliplatin 85 mg/m², d1 every two weeks (q2w) 4 cycles (8 weeks) pre-OP and 4 cycles (8 weeks) post-OP
  Interventions: Drug: Docetaxel; Drug: Oxaliplatin; Drug: Leucovorin; Drug: Fluorouracil

INTERVENTIONS:
Drug: Docetaxel — 50mg/m2, d1, i.v., every 2 weeks
  Arms: Perioperative FLOT chemotherapy
Drug: Oxaliplatin — 85 mg/m², d1, i.v., every 2 weeks
  Arms: Perioperative FLOT chemotherapy
Drug: Leucovorin — 200 mg/m², d1, i.v., every 2 weeks
  Arms: Perioperative FLOT chemotherapy
Drug: Fluorouracil — 2600 mg/m²d1 i.v. every 2 weeks
  Arms: Perioperative FLOT chemotherapy
Drug: Capecitabine — 1000 mg/m² two times per day (BID), d1-14
  Arms: Perioperative XELOX chemotherapy
Drug: Oxaliplatin — 130 mg/m² d1 i.v. every 3 weeks
  Other Names: oxaliplatine
  Arms: Perioperative XELOX chemotherapy

SUMMARY:
Patients with resectable adenocarcinoma of stomach or esophagogastric junction without previous therapy will be treated with one of two chemotherapy regimens perioperatively. One group of the patients will receive 5-Fluorouracil (5-FU), Leucovorin, Oxaliplatin and Docetaxel (FLOT), the second group will receive Oxaliplatin and Capecitabin (XELOX). Primary endpoint of the study is the proportion of patients who complete all allocated treatment.

DETAILED DESCRIPTION:
328 рatients with resectable (T1b-4 and/or N-/+, M0) adenocarcinoma of the stomach or the esophagogastric junction without previous therapy will be included in this study. After staging laparocopy patients will be randomized to receive preoperatively 4 cycles FLOT or 4 cycles XELOX followed by curative surgery. Adjuvant chemotherapy will be given as 4 cycles of FLOT or 4 cycles XELOX. The primary endpoint is the proportion of patients who fully adhered to all the allocated treatment per protocol. Secondary endpoints are pathological regression grade, progression free survival, overall survival, chemotherapy and surgery complications rates.

ELIGIBILITY:
Inclusion Criteria:

* cT1b-T4b (cT4b - invasion in diaphragm, parenchyma of liver, spleen, pancreas, abdominal wall, small bowel, colon, distal part of splenic artery)
* cN0-3
* M0
* Age: 18 - 80
* ECOG: 0 - 1
* Histological type: adenocarcinoma
* Differentiation grade: G0 - G4
* No previous surgery
* No previous chemotherapy
* No concomitant severe comorbidity
* Written informed consent

Exclusion Criteria:

* cT1a, cT4b (invasion in truncus, hepatic artery, proximal part of splenic artery)
* Presense of distant metastases
* ECOG: 2 - 5
* Age: <18 and >80
* Severe concomitant comorbidity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who complete all the treatment per protocol | Up to 2 months
  Completed treatment protocol is considered as 4 cycles neoadjuvant chemotherapy followed by curative surgery and 4 cycles of adjuvant chemotherapy.

SECONDARY OUTCOMES:
Chemotherapy toxicity profile | at the end of XELOX cycle (each cycle is 21 days) and FLOT cycle (each cycle is 14 days)
  To determine and compare toxicity profile in patients receiving XELOX or FLOT regimen
Surgical complications rate | up to 90th day after surgery
  To determine surgical complication rate and profile after different types of regimens in neoadjuvant settings
1-year disease-free survival rate | 1 year after surgery
  To determine the efficacy of FLOT regimen compared to XELOX regimen during the first year after the surgery
Correlation between histopathological regression and disease-free survival | 2 years of follow-up after the last cycle of chemotherapy
  To determine correlation between histopathological regression and disease-free survival in different chemotherapeutic settings
Median overall survival | 5 year follow up after the last cycle of chemotherapy
  To determine the efficacy of FLOT regimen compared to XELOX regimen by assessment of overall survival
Histopathological regression rate (Becker regression criteria) | 2 weeks after surgery
  To determine histopathological regression rate after FLOT regimen compared to XELOX regimen in neoadjuvant settings

CONTACTS AND LOCATIONS:
Overall Officials: Oleksii Dobrzhanskyi, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: Yes
After the initial publication every participant will recieve all the data to provide further data exploration.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available after initial paper is published.
Access Criteria: By request

REFERENCES:
- [Derived] Dobrzhanskyi O, Kopetskyi V, Ross EA, Chernoff J, Shudrak Y, Kolesnyk A, Pepenin M, Horodetskyi A, Melnitchouk N, Kondratskyi Y. Treatment discontinuation associated with perioperative toxicity of FLOT versus XELOX chemotherapy in patients with resectable gastric cancer: prospective randomized trial (PECORINO). J Gastrointest Oncol. 2025 Jun 30;16(3):909-921. doi: 10.21037/jgo-2024-921. Epub 2025 Jun 24. PMID 40672074